CLINICAL TRIAL: NCT03373409
Title: An Open-label, Single-Center, Single-Dose, 3-Way Crossover Study of the Safety and Pharmacokinetics of Albuterol Administered by the Halix(TM) Albuterol Unit Dose Disposable Inhaler
Brief Title: Safety and Pharmacokinetics of Halix(TM) Albuterol Unit Dose Disposable Inhaler Versus Albuterol MDI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Concentrx Pharmaceuticals, Inc. (Industry)
Collaborators: PharPoint Research, Inc. (Industry); Kramer Consulting, LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CONX-101
Record Dates: First submitted 2017-10-03; First posted 2017-12-14 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Asthma
Keywords: Dry Powder Inhaler
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: 3-way single dose crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Albuterol DPI 90mcg (Experimental): Participants will receive albuterol 90mcg via the albuterol DPI
  Interventions: Drug: Albuterol DPI 90mcg
- Albuterol DPI 180mcg (Experimental): Participants will receive albuterol 180mcg via the albuterol DPI
  Interventions: Drug: Albuterol DPI 180mcg
- Albuterol HFA MDI (Active Comparator): Participants will receive albuterol 180mcg via the HFA MDI inhaler
  Interventions: Drug: Albuterol HFA MDI

INTERVENTIONS:
Drug: Albuterol DPI 90mcg — Albuterol unit dose disposable DPI delivers 90mcg of albuterol in the excipient lactose with each inhalation. Albuterol 90mcg will be given on one of the 3 treatment days. One inhalation from the DPI will be used.
  Other Names: Halix (TM) albuterol unit dose disposable inhaler
  Arms: Albuterol DPI 90mcg
Drug: Albuterol DPI 180mcg — Albuterol unit dose disposable DPI delivers 90mcg of albuterol in the excipient lactose with each inhalation. Albuterol 180mcg will be given on one of the 3 treatment days. Two inhalations from the DPI will be used to deliver the 180mcg dose
  Other Names: Halix (TM) albuterol unit dose disposable inhaler
  Arms: Albuterol DPI 180mcg
Drug: Albuterol HFA MDI — Albuterol HFA MDI delivers 90mcg of albuterol with each inhalation. Albuterol 180mcg will be given on one of the 3 treatment days. Two inhalations from the MDI will be used to deliver the 180mcg dose
  Other Names: Ventolin HFA MDI
  Arms: Albuterol HFA MDI

SUMMARY:
Healthy male and female volunteers without asthma will be recruited to enroll in a single dose 3-way crossover study of the safety and pharmacokinetics of albuterol when administered using the Halix (TM) albuterol unit dose disposable dry powder inhaler (DPI) and the albuterol HFA (hydrofluoroalkane) MDI inhaler.

DETAILED DESCRIPTION:
The study objective is to compare the safety of albuterol in a dry powder inhaler (DPI) and albuterol in an HFA metered dose inhaler (MDI) after single albuterol doses of 90mcg and 180mcg delivered by the DPI and 180mcg delivered by the MDI. Another study objective is to compare the pharmacokinetics (metabolism) of albuterol with the two inhalers in all subjects treated. To participate in the study, subjects must provide written informed consent, washout any prohibited medications and pass all the screening criteria. Once this is done, there will be 3 treatment visits for each subject. At each of these visits, the subject will inhale from either the DPI or the MDI. Assignment of subjects to one of six (6) unique sequences of treatment will be according to a randomized scheme. The subject will inhale albuterol either once from the DPI (90mcg), twice from the DPI (180mcg) and twice from the MDI (180mcg). Following inhalation of the study drug, there will be a series of assessments taken at times postdose with spirometry (FEV1) measured up to 2 hours postdose, vital signs measured up to 10 hours post dose, ECGs obtained up to 5 hours postdose, blood taken to measure potassium and glucose up to 6 hours postdose, and blood for pharmacokinetic evaluation obtained up to 10 hours postdose. A washout period of 60 to 192 hours will separate each of the 3 treatment visits. Following these visits, there will be a study concluding visit 3 to 10 days later.

ELIGIBILITY:
Inclusion Criteria:Subjects are required to meet ALL of the following inclusion criteria to be eligible for enrollment in the study.

1. Has provided written informed consent
2. Speaks and understands the English language
3. Males or females 18 to 55 years of age (inclusive) at the Consent Visit
4. Nonsmoker or ex-smoker who has abstained from smoking for at least 1 year prior to the Consent Visit and who has a ≤ 15 pack/year history of lifetime cigarette use
5. Has no history of use of nicotine gum, nicotine patch, e-cigarettes/vaping preparations in the 3 months before the Consent Visit
6. Has a body mass index (BMI) of 18.5 to 35.0 (calculated as kg/m2)
7. Has never had a diagnosis of asthma, exercise-induced bronchospasm, chronic obstructive pulmonary disease, or other chronic respiratory disease or chronic upper airway condition (seasonal or perennial allergic rhinitis is not exclusionary; however, nasal polypectomy within the 12 months prior to the Screening Visit is exclusionary
8. Has a FEV1 ≥ 80% of predicted normal for age, gender, height and ethnicity (percent of predicted normal values for FEV1 will be calculated using National Health and Nutrition Examination Survey III [NHANES III]) calculation at the Screening Visit
9. Has a FEV1/FVC ratio ≥ 0.70 at the Screening Visit
10. Ability to maintain a peak inspiratory flow rate of at least 60 L/min measured by the In-check DIAL device at the medium resistance setting.
11. At the Screening Visit, demonstrates adequate understanding of and ability to successfully inhale from an MDI as determined by the investigator and through demonstrated successful use of the Vitalograph® aerosol inhalation monitor (AIM™) (training/validation device for MDI) using a placebo MDI canister.

[Note: potential subjects who cannot demonstrate successful MDI technique using with the AIM device (with placebo canister) after in-clinic training at the Screening Visit will not be eligible for continued participation in the study.] 12. At the Screening Visit, demonstrates adequate understanding of and ability to successfully inhale when using the Halix™ UDDI [Note: a placebo UDDI not containing any drug powder will be supplied for each potential subject to become familiar with the inhaler and practice inhalation technique] [Note: potential subjects who cannot demonstrate successful inhalation technique using the Halix™ UDDI after in-clinic training at the Screening Visit will not be eligible for continued participation in the study].

13. Willing and able to comply with all aspects of the study protocol including avoiding use of certain concomitant medications and attending the required clinic visits (ie, has no conflicting plans that would prohibit attendance at scheduled study visits including each of the threeTreatment Day Visits)

-

Exclusion Criteria:Subjects will be excluded from participation in the study if ANY of the following criteria are present:

1. Female subjects of childbearing potential (CBP) who are not using reliable contraception (eg, abstinence, double barrier method, oral/implantable/transdermal contraception, Depo-Provera, intrauterine device); a woman is of CBP unless she is premenarchal, is at least 2 years postmenopausal, is without a uterus and/or both ovaries, has had a bilateral tubal ligation, or has undergone the Essure procedure with confirmation of tubal blockage.

   [Note: If a female is identified as less than 2 years postmenopausal, a serum follicle-stimulating hormone (FSH) determination will be performed as a part of screening laboratory assessments. If a FSH result of < 40 mIU/mL is obtained, the female will be determined to be of CBP and her unwillingness to use reliable contraception as defined above will be exclusionary for the study.]
2. A woman who is pregnant (has a positive serum pregnancy test at Screening), is lactating, or is likely/planning to become pregnant during the study
3. Vital signs at the Screening Visit (after at least 2 minutes seated at rest) showing SBP either < 80 mmHg or >150 mmHg; DBP > 90 mmHg; or HR either < 40 bpm or > 100 bpm (vital signs outside these criteria may be repeated once after an additional seated rest period of at least 2 minutes- if vital signs exclusion criteria are not met after the repeat measurements of SBP, DBP, or HR, screening may continue)
4. Emergency room visit or hospitalization for any acute respiratory condition in the 3 months prior to the Screening Visit
5. Currently receiving pharmacologic treatment for diabetes or hypertension
6. History of any acute or chronic hepatobiliary disorder or documented elevation of alanine transaminase (ALT) or aspartate transaminase (AST) 2 or more times the upper limit of the normal (ULN) laboratory reference range in the 12 months prior to the Consent Visit,
7. Clinical laboratory results (after ≥4 hours fasting) at the Screening Visit that show any one or more of the following:

   * hemoglobin < 13.5 g/dL in male subjects; < 12 g/dL in female subjects
   * hematocrit < 38 % in male subjects; <35% in female subjects
   * total white blood cell count (WBC) < 2500 cells/mm3
   * platelet count < 150,000 cells/mm3
   * serum glucose < 80 mg/dL or > 120 mg/dL
   * serum potassium < 3.5 mmol/L or > 5.2 mmol/L
   * ALT or AST > 2.0 times ULN
   * alkaline phosphatase (ALP) > 1.5 times ULN
   * serum creatinine > 1.5 times ULN
   * positive serum hCG (female subjects only)
   * positive serologic test for HBsAg, anti-HCV antibody, or HIV antibody
   * in the opinion of the investigator, a urinalysis result showing medically significant abnormality
   * positive urine drug screen [Exception: urine drug screen detects evidence of an authorized prescribed medication]
   * positive urine cotinine test
8. Presence of any uncontrolled (in the Investigator's medical opinion) systemic disease, including, but not limited to renal, hepatic, hematologic, gastrointestinal, endocrine, pulmonary, cardiac, neurologic, or psychiatric disease
9. Electrocardiogram obtained at Screening Visit that shows medically significant abnormalities (e.g., left bundle branch block, frequent premature ventricular contractions, chronic atrial fibrillation, or QTc interval prolongation > 450 msec for males and > 470 msec for females)
10. Has a FEV1 < 80% of that predicted for age, gender, height, and ethnicity at the Screening Visit based on NHANES III calculation.
11. Has a FEV1 / FVC ratio < 0.70
12. Inability to maintain a peak inspiratory flow rate of 60 L/min or higher
13. Presence of a current condition (e.g., alcoholism [or consumption of substantial quantities of alcohol], drug abuse, or psychiatric condition) making it unlikely that the requirements of the subject's participation in the protocol will be met
14. History of allergic reaction (known hypersensitivity) to albuterol sulfate and/or lactose, in any formulation, or history of severe hypersensitivity to milk proteins
15. Current participation in a drug, drug/device or biologic investigational research study or participation in a drug, drug/device or biologic investigational research study within the 30 days prior to the Screening Visit
16. An elective surgical or medical procedure currently is planned or scheduled to be performed during the study (this excludes routine immunotherapy/desensitization procedures that are being performed on a regular schedule and have been unchanged for at least 3 months prior to the Screening Visit)
17. Presence of a clinically diagnosed upper respiratory tract infection within the 14 days prior to the Screening Visit
18. Has undergone nasal polypectomy within the 12 months prior to the Screening Visit

    -

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2018-05-28 (Actual); Study Completion 2018-07-25 (Actual)

PRIMARY OUTCOMES:
Forced Expiratory Volume in 1 second (FEV1) before and after oral inhalation of albuterol on 3 different treatment days | At each of the 3 treatment visits, FEV1 (forced expiratory volume in one second) will be measured prior to drug administration and 6 times after dose- at 5 min, 15 min, 30 min, 45 min, 60 min and 120 min.
  Change from treatment day baseline in forced expiratory volume in one second (FEV1) will be assessed serially up to 120 minutes after each of 3 single doses of inhaled albuterol

SECONDARY OUTCOMES:
Systolic and diastolic blood pressure before and after oral inhalation of albuterol on 3 different treatement days | Serial measurements of systolic and diastolic blood pressure will be taken at baseline (15-40 mnutes pre-dose) and at 15, 30, 45, 60, 120 minutes post dose and at 3, 4, 5, 6, 10, 12, and 14 hours post-dose
  Change from treatment day baseline in blood pressure will be evaluated by the maximum change (systolic) and minimum change (diastolic) from baseline blood pressure, and the weighted mean change form baseline in systolic and diastolic blood pressure
Serum potassium before and after oral inhalation of albuterol on 3 different treatment days | Serial measurments of serum potassium will be obtained at 10, 20, 30, 45, 60 and 120 minutes post-dose and 3 and 4 hours post-dose
  Change from treatment day baseline in serum potassium after each of 3 single doses of inhaled albuterol will be evaluated by the description of change from baseline values
Serum glucose before and after oral inhalation of albuterol on 3 different treatment days | Serial measurments of serum potassium will be obtained at 10, 20, 30, 45, 60 and 120 minutes post-dose and 3 and 4 hours post-dose
  Change from treatment day baseline in serum glucose after each of 3 single doses of inhaled albuterol will be evaluated by the description of change from baseline values
Electrocardiographic QTc interval before and after oral inhalation of albuterol on 3 different treatment days | Serial ECGs (electrocardiograms) will be taken at baseline (5-40 minutes pre-dose), 10 min post-dose, 50 min post-dose, and 5 hours post-dose.
  Change from treatment day baseline ECG (electrocardiogram) will assess the maximum and mean change from baseline of the corrected QT interval (QT measures the time between the start of the Q wave and the end of the T wave in the heart's electrical cycle) following each of the 3 single doses of inhaled albuterol study drug.

OTHER OUTCOMES:
Peak plasma concentration (Cmax) of albuterol after oral inhalation on 3 different treatment days | PK samples to be collected postdose at 5, 10, 20, 30, 45, 60, and 120 minutes, and at 3, 4, 5, 6, 10, 12, and 14 hours post-dose
  Predose and post dose measurement of albuterol in plasma will be assessed after each of 3 single doses of inhaled albuterol.
Area under the plasma concentration versus time (AUC0-t) of albuterol after oral inhalation on 3 different treatment days | PK samples to be collected postdose at 5, 10, 20, 30, 45, 60, and 120 minutes, and at 3, 4, 5, 6, 10, 12, and 14 hours post-dose
  Predose and post dose measurement of albuterol in plasma will be assessed after each of 3 single doses of inhaled albuterol.
Area under the plasma concentration versus time to infinity (AUC0-inf) of albuterol after oral inhalation on 3 different treatment days | PK samples to be collected postdose at 5, 10, 20, 30, 45, 60, and 120 minutes, and at 3, 4, 5, 6, 10, 12, and 14 hours post-dose
  Predose and post dose measurement of albuterol in plasma will be assessed after each of 3 single doses of inhaled albuterol.
Time to maximum plasma concentration (tmax) of albuterol after oral inhalation on 3 different treatment days | PK samples to be collected postdose at 5, 10, 20, 30, 45, 60, and 120 minutes, and at 3, 4, 5, 6, 10, 12, and 14 hours post-dose
  Predose and post dose measurement of albuterol in plasma will be assessed after each of 3 single doses of inhaled albuterol.
Apparent terminal half-life (t 1/2) of albuterol after oral inhalation on 3 different treatment days | PK samples to be collected postdose at 5, 10, 20, 30, 45, 60, and 120 minutes, and at 3, 4, 5, 6, 10, 12, and 14 hours post-dose
  Predose and post dose measurement of albuterol in plasma will be assessed after each of 3 single doses of inhaled albuterol.
Estimation of the terminal elimination rate constant (lambda z) of albuterol after oral inhalation on 3 different treatment days | PK samples to be collected postdose at 5, 10, 20, 30, 45, 60, and 120 minutes, and at 3, 4, 5, 6, 10, 12, and 14 hours post-dose
  Predose and post dose measurement of albuterol in plasma will be assessed after each of 3 single doses of inhaled albuterol.

CONTACTS AND LOCATIONS:
Overall Officials: William J Alexander, MD, Study Chair — Concentrx Pharmaceuticals
Locations (1):
- North Carolina Clinical Research, Raleigh, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No